CLINICAL TRIAL: NCT05592938
Title: Partial Breast Re-irradiation Using Ultra Hypofractionation: Phase 2 Multi-institutional Study (PRESERVE)
Brief Title: Partial Breast Re-irradiation Using Ultra Hypofractionation (PRESERVE)
Acronym: PRESERVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Royal Victoria Regional Health Centre (Unknown); AC Camargo Cancer Center (Other); King Hussein Cancer Center (Other); Tata Memorial Hospital (Other Government); NYU Langone Health (Other); Centre hospitalier de l'Université de Montréal (CHUM) (Other); Peter MacCallum Cancer Centre, Australia (Other); CHU de Quebec-Universite Laval (Other); l'Hopital Maisonneuve-Rosemont (Unknown); L'Institut de recherche du Centre universitaire de sante McGill (Unknown); Florence University Hospital (Unknown); Tel-Aviv Sourasky Medical Center (Other Government); Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-5074
Record Dates: First submitted 2022-10-14; First posted 2022-10-25 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer; Breast Cancer Recurrent
Keywords: Hypofractionated
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- rPBI (Experimental): 26Gy in 5 daily fractions over 1-week
  Interventions: Radiation: rPBI

INTERVENTIONS:
Radiation: rPBI — External beam partial breast reirradiation (rPBI) using 26Gy in 5 fractions delivered daily over 1-week

SUMMARY:
Breast-conserving surgery followed by re-irradiation with partial breast irradiation (rPBI) has recently been found to be a safe alternative to mastectomy for women who have undergone prior whole breast radiation. By reducing the volume of tissue receiving radiation, rPBI has been associated with less toxicity and improved cosmetic outcomes. For many women with early-stage breast cancer, shorter 1-week (5-fraction) courses of breast radiation (ultra-fractionation) have been found to be equivalent to longer fractionation schedules in the upfront treatment setting. These 1-week schedules are more convenient for patients, with fewer treatments and shorter overall treatment time. The investigators hypothesize that a 1-week ultra-hypofractionated rPBI regimen following breast-conserving surgery (BCS) for local recurrence or new primary breast cancer in the previously irradiated breast (LR) will be associated with acceptable toxicity at 1 year (<13% grade >3 toxicity).

DETAILED DESCRIPTION:
Most women affected by breast cancer are treated with breast-conserving surgery to remove the tumour, followed by radiation to reduce the risk of recurrence. Unfortunately, some women will experience recurrence of the cancer in the previously treated breast. These recurrences have historically been treated by removing the whole breast or a second breast-conserving surgery followed by 3 to 5 weeks of radiation. These treatments can negatively impact mental health and quality of life or lead to harmful side effects that could impact the skin, breast, ribs, heart and lungs.

Breast-conserving surgery followed by re-irradiation with partial breast irradiation (rPBI) has recently been found to be a safe alternative to mastectomy for women who have undergone prior whole breast radiation. By reducing the volume of tissue receiving radiation, rPBI has been associated with less toxicity and improved cosmetic outcomes. For many women with early-stage breast cancer, shorter 1-week (5-fraction) courses of breast radiation (ultra-fractionation) have been found to be equivalent to longer fractionation schedules in the upfront treatment setting. These 1-week schedules are more convenient for patients, with fewer treatments and shorter overall treatment time. The investigators hypothesize that a 1-week ultra-hypofractionated rPBI regimen following breast-conserving surgery (BCS) for local recurrence or new primary breast cancer in the previously irradiated breast (LR) will be associated with acceptable toxicity at 1 year (<13% grade >3 toxicity).

The target population for this study is women with localized recurrent or new primary breast cancer in the previously irradiated breast. This is a prospective single arm phase 2 trial of external beam rPBI using 26Gy in 5 fractions delivered daily over 1-week after a second lumpectomy for LR following prior BCS and adjuvant whole or partial breast irradiation. Using a multi-institutional and international network of comprehensive cancer centers, this study will advance global knowledge of how to optimally treat women with this disease.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* In-breast recurrence or new primary (ductal carcinoma in situ (DCIS) or invasive carcinoma)
* Tumour <3.0 cm in greatest diameter on pathologic examination, including both invasive and non-invasive components
* >5 years after completion of prior adjuvant whole or partial breast radiotherapy (prior nodal radiotherapy permitted)
* Clinically node negative
* Negative margins (no tumour on ink)
* Recovered from surgery with the incision completely healed and no signs of infection

Exclusion Criteria:

* Multicentric disease (patients with multifocal breast cancer in the same quadrant are eligible)
* Tumour histology limited to lobular carcinoma only
* Extensive intraductal component
* T4 disease
* Node positive or distant metastatic disease
* Serious non-malignant disease (cardiovascular, pulmonary, systemic lupus erythematosus, scleroderma), which would preclude radiation treatment
* Currently pregnant or lactating
* Presence of an ipsilateral breast implant or pacemaker
* Unable to commence radiation within 16 weeks of breast-conserving surgery (or last surgical procedure on the breast) or within 12 weeks from last cycle of adjuvant chemotherapy
* Unable to clearly define the surgical cavity (oncoplastic procedures are permitted provided the tumor bed is well delineated with surgical clips).
* Psychiatric disorders which would preclude obtaining informed consent or adherence to protocol
* Grade II or more late skin toxicity from prior radiation evaluated and graded using CTCAE v5.0

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2027-06-27 (Estimated); Study Completion 2027-06-27 (Estimated)

PRIMARY OUTCOMES:
Grade ≥3 toxicity associated with treatment | During accrual period, up to 3 years
  TThe primary endpoint, grade ≥3 toxicity associated with treatment will be summarized using frequency and percentage with 95% Clopper-Pearson confidence intervals by grade at each scheduled follow up.

SECONDARY OUTCOMES:
Frequency radiation-associated toxicity (acute) | 3 months, 1 year, 2 year, 3 years, 4 years and 5 years post rPBI
  Radiation-associated toxicities (acute) will be graded according to CTCAE v5.0 by physicians. Toxicity associated with treatment will be summarized using frequency with 95% Clopper-Pearson confidence intervals by grade at each scheduled follow up.
Percentage radiation-associated toxicity (acute) | 3 months, 1 year, 2 year, 3 years, 4 years and 5 years post rPBI
  Radiation-associated toxicities (acute) will be graded according to CTCAE v5.0 by physicians. Toxicity associated with treatment will be summarized using percentage with 95% Clopper-Pearson confidence intervals by grade at each scheduled follow up.
Frequency radiation-associated toxicity (late) | 3 months, 1 year, 2 year, 3 years, 4 years and 5 years post rPBI
  Radiation-associated toxicities (late) will be graded according to CTCAE v5.0 by physicians. Toxicity associated with treatment will be summarized using frequency with 95% Clopper-Pearson confidence intervals by grade at each scheduled follow up.
Percentage radiation-associated toxicity (late) | 3 months, 1 year, 2 year, 3 years, 4 years and 5 years post rPBI
  Radiation-associated toxicities (late) will be graded according to CTCAE v5.0 by physicians. Toxicity associated with treatment will be summarized using percentage with 95% Clopper-Pearson confidence intervals by grade at each scheduled follow up.
Risk of local recurrence (invasive and DCIS) | 3 months, 1 year, 2 year, 3 years, 4 years and 5 years post rPBI
  Cumulative incidence function will be used to estimate local recurrence with death as a competing risk.
Risk of distant recurrence (invasive and DCIS) | 3 months, 1 year, 2 year, 3 years, 4 years and 5 years post rPBI
  Cumulative incidence function will be used to estimate distant recurrence and distance recurrence with death as a competing risk.
Location of local recurrence (in-field) (frequency) | 3 months, 1 year, 2 year, 3 years, 4 years and 5 years post rPBI
  Location of recurrence will be summarized by frequency.
Location of local recurrence (in-field) (percentage) | 3 months, 1 year, 2 year, 3 years, 4 years and 5 years post rPBI
  Location of recurrence will be summarized by percentage.
Location of local recurrence (out-of-field) (frequency) | 3 months, 1 year, 2 year, 3 years, 4 years and 5 years post rPBI
  Location of recurrence will be summarized by frequency.
Location of local recurrence (out-of-field) (percentage) | 3 months, 1 year, 2 year, 3 years, 4 years and 5 years post rPBI
  Location of recurrence will be summarized by percentage
Risk of local recurrence after rPBI requiring mastectomy | 3 months, 1 year, 2 year, 3 years, 4 years and 5 years post rPBI
  Cumulative incidence function will be used to estimate local recurrence after rPBI requiring mastectomy with death as a competing risk
Invasive breast cancer free survival | 3 months, 1 year, 2 year, 3 years, 4 years and 5 years post rPBI
  Kaplan-Meier method will be used to estimate invasive breast cancer free survival
Overall survival | 3 months, 1 year, 2 year, 3 years, 4 years and 5 years post rPBI
  Kaplan-Meier method will be used to estimate overall survival
Satisfaction with breasts | Baseline, 1 year, 3 years, and 5 years post rPBI
  Quality of life questionnaire will be used to obtain scores and will summarized using mean and standard deviation at baseline and follow up. Change in score compared to baseline will be summarized using mean and standard deviation, and assessed with paired t-test. Number and proportion of patients with a minimal clinically important difference will be calculated.
Financial toxicity associated with treatment | Baseline, 3 months, 1 year, and 3 years post rPBI
  Quality of life questionnaire will be used to obtain scores and will summarized using mean and standard deviation at baseline and follow up. Change in score compared to baseline will be summarized using mean and standard deviation, and assessed with paired t-test. Number and proportion of patients with a minimal clinically important difference will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Rodin, MD, Principal Investigator — Princess Margaret Cancer Centre; Anne Koch, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (15):
- United States (3):
  - NYU Langone Health, New York, New York
  - Columbia University Medical Center, New York, New York
  - Virgina Community University Massey Comprehensive Cancer Center, Richmond, Virginia
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia
- A.C.Camargo Cancer Center, São Paulo, São Paulo, Brazil
- Canada (7):
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Verspeeten Family Cancer Centre, London, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - CHU de Québec-Université Laval, Montreal, Quebec
  - Hôpital Maisonneuve-Rosemont - CIUSSS de l'Est-de-l'Île-de-Montréal, Montreal, Quebec
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
- Tel-Aviv Sourasky Medical Centre, Tel Aviv, Israel
- Florence University Hospital, Florence, Italy
- King Hussein Cancer Centre, Amman, Jordan, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Loibl S, Poortmans P, Morrow M, Denkert C, Curigliano G. Breast cancer. Lancet. 2021 May 8;397(10286):1750-1769. doi: 10.1016/S0140-6736(20)32381-3. Epub 2021 Apr 1. PMID 33812473
- [Background] Fingeret MC, Nipomnick S, Guindani M, Baumann D, Hanasono M, Crosby M. Body image screening for cancer patients undergoing reconstructive surgery. Psychooncology. 2014 Aug;23(8):898-905. doi: 10.1002/pon.3491. Epub 2014 Feb 6. PMID 25066586
- [Background] Martei YM, Vanderpuye V, Jones BA. Fear of Mastectomy Associated with Delayed Breast Cancer Presentation Among Ghanaian Women. Oncologist. 2018 Dec;23(12):1446-1452. doi: 10.1634/theoncologist.2017-0409. Epub 2018 Jun 29. PMID 29959283
- [Background] Arthur DW, Winter KA, Kuerer HM, Haffty B, Cuttino L, Todor DA, Anne PR, Anderson P, Woodward WA, McCormick B, Cheston S, Sahijdak WM, Canaday D, Brown DR, Currey A, Fisher CM, Jagsi R, Moughan J, White JR. Effectiveness of Breast-Conserving Surgery and 3-Dimensional Conformal Partial Breast Reirradiation for Recurrence of Breast Cancer in the Ipsilateral Breast: The NRG Oncology/RTOG 1014 Phase 2 Clinical Trial. JAMA Oncol. 2020 Jan 1;6(1):75-82. doi: 10.1001/jamaoncol.2019.4320. PMID 31750868
- [Background] Korzets Y, Lee G, Espin-Garcia O, Purdie T, Koch AC, Hodgson D, Barry A, Fyles A. The Role of Partial Breast Radiation in the Previously Radiated Breast. Am J Clin Oncol. 2019 Dec;42(12):932-936. doi: 10.1097/COC.0000000000000584. PMID 31436745
- [Background] Brunt AM, Haviland JS, Sydenham M, Agrawal RK, Algurafi H, Alhasso A, Barrett-Lee P, Bliss P, Bloomfield D, Bowen J, Donovan E, Goodman A, Harnett A, Hogg M, Kumar S, Passant H, Quigley M, Sherwin L, Stewart A, Syndikus I, Tremlett J, Tsang Y, Venables K, Wheatley D, Bliss JM, Yarnold JR. Ten-Year Results of FAST: A Randomized Controlled Trial of 5-Fraction Whole-Breast Radiotherapy for Early Breast Cancer. J Clin Oncol. 2020 Oct 1;38(28):3261-3272. doi: 10.1200/JCO.19.02750. Epub 2020 Jul 14. PMID 32663119
- [Background] Murray Brunt A, Haviland JS, Wheatley DA, Sydenham MA, Alhasso A, Bloomfield DJ, Chan C, Churn M, Cleator S, Coles CE, Goodman A, Harnett A, Hopwood P, Kirby AM, Kirwan CC, Morris C, Nabi Z, Sawyer E, Somaiah N, Stones L, Syndikus I, Bliss JM, Yarnold JR; FAST-Forward Trial Management Group. Hypofractionated breast radiotherapy for 1 week versus 3 weeks (FAST-Forward): 5-year efficacy and late normal tissue effects results from a multicentre, non-inferiority, randomised, phase 3 trial. Lancet. 2020 May 23;395(10237):1613-1626. doi: 10.1016/S0140-6736(20)30932-6. Epub 2020 Apr 28. PMID 32580883
- [Background] Barrios CH, Reinert T, Werutsky G. Global Breast Cancer Research: Moving Forward. Am Soc Clin Oncol Educ Book. 2018 May 23;38:441-450. doi: 10.1200/EDBK_209183. PMID 30231347
- [Background] Abdel-Razeq H, Mansour A, Jaddan D. Breast Cancer Care in Jordan. JCO Glob Oncol. 2020 Feb;6:260-268. doi: 10.1200/JGO.19.00279. PMID 32083950
- [Background] Khader J, Glicksman RM, Mheid S, Mansour A, Giuliani ME, Gospodarowicz M, Almousa A, Abdel-Razeq H, Rodin D. Enhancing International Cancer Organization Collaborations: King Hussein Cancer Center and Princess Margaret Cancer Centre Model for Collaboration. J Cancer Educ. 2022 Jun;37(3):763-769. doi: 10.1007/s13187-020-01878-z. Epub 2020 Sep 14. PMID 32926325
- [Background] Rodin D, Tawk B, Mohamad O, Grover S, Moraes FY, Yap ML, Zubizarreta E, Lievens Y. Hypofractionated radiotherapy in the real-world setting: An international ESTRO-GIRO survey. Radiother Oncol. 2021 Apr;157:32-39. doi: 10.1016/j.radonc.2021.01.003. Epub 2021 Jan 14. PMID 33453312